CLINICAL TRIAL: NCT00372502
Title: Lactate Assessment in the Treatment of Early Sepsis: The LactATES Trial
Brief Title: Clinical Trial of the Optimal Endpoint of Early Sepsis Resuscitation
Acronym: LactATES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Alan E Jones, MD; Assistant Research Director, Carolinas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1K23GM076652 (NIH)
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: sepsis; shock; emergency department; resuscitation
MeSH Terms: conditions — Sepsis; Shock, Septic; Shock; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Procedure: Standard EGDT
- 2 (Experimental)
  Interventions: Procedure: Modified EGDT

INTERVENTIONS:
Procedure: Modified EGDT — Early goal directed therapy with lactate clearance
  Arms: 2
Procedure: Standard EGDT — Early goal directed therapy
  Arms: 1

SUMMARY:
The purpose of this study is to determine if there is equivalence between two different methods of treating patients with severe bloodstream infection called sepsis. We will randomly assign patients to one of two treatment methods. One of the treatment methods is the current standard of care and uses an infrared sensor on the end of a catheter to determine the adequacy of treatment. The second treatment method is identical to the first but instead of the infrared sensor a blood test that is performed as a part of standard care (with blood drawn from the catheter) will be used to determine the adequacy of treatment. This study will attempt to determine an easier method of guiding treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected infection
2. Any two of four criteria of systemic inflammatory response
3. SBP < 90 mm Hg after 20cc/kg crystalloid (septic shock) or either a whole blood lactate > 4 mmol/L (severe sepsis).

Exclusion Criteria:

1. Age < 18 years
2. Pregnancy
3. Established "Do Not Resuscitate" orders prior to enrollment
4. Primary diagnosis other than sepsis
5. Requirement for immediate surgery in < 6 hours from admission
6. Any absolute contraindication to central venous catheterization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Mortality | In-hospital

CONTACTS AND LOCATIONS:
Overall Officials: Alan E Jones, MD, Study Director — Carolinas Medical Center; Jeffrey A Kline, MD, Study Chair — Carolinas Medical Center
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Cooper Hospital, Camden, New Jersey
  - Carolinas Medical Center, Charlotte, North Carolina

REFERENCES:
- [Derived] Puskarich MA, Trzeciak S, Shapiro NI, Albers AB, Heffner AC, Kline JA, Jones AE. Whole blood lactate kinetics in patients undergoing quantitative resuscitation for severe sepsis and septic shock. Chest. 2013 Jun;143(6):1548-1553. doi: 10.1378/chest.12-0878. PMID 23740148
- [Derived] Jones AE, Shapiro NI, Trzeciak S, Arnold RC, Claremont HA, Kline JA; Emergency Medicine Shock Research Network (EMShockNet) Investigators. Lactate clearance vs central venous oxygen saturation as goals of early sepsis therapy: a randomized clinical trial. JAMA. 2010 Feb 24;303(8):739-46. doi: 10.1001/jama.2010.158. PMID 20179283